CLINICAL TRIAL: NCT05141864
Title: Acmella Oleracea in the Analgesia of the Digital Rectal Examination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Fabrizia Serra Pereira Guerrieri, Principal investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Acmella
Record Dates: First submitted 2021-11-20; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Analgesia in the Digital Rectal Examination
Keywords: Prostatic neoplasms; Digital Rectal Examination; Phytotherapy; Pain; Analgesia; Spilanthes oleracea
MeSH Terms: conditions — Prostatic Neoplasms; Pain; Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acmella oleracea gel group (Active Comparator): Formulation with Acmella oleracea will be used during the digital rectal examination.
  Interventions: Biological: Acmella oleracea gel
- Lidocaina gel group (Active Comparator): The lidocaine gel will be used during the digital rectal examination.
  Interventions: Drug: Lidocaine 2 % Topical Cream
- Ultrasound gel group (Placebo Comparator): The ultrasound gel will be used during the digital rectal examination.
  Interventions: Other: Ultrasound gel

INTERVENTIONS:
Biological: Acmella oleracea gel — Study group will use Acmella oleracea gel during the digital rectal examination.
  Arms: Acmella oleracea gel group
Drug: Lidocaine 2 % Topical Cream — Control group will use lidocaine 2% gel during the digital rectal examination.
  Arms: Lidocaina gel group
Other: Ultrasound gel — Control group will use ultrasound gel during the digital rectal examination.
  Arms: Ultrasound gel group

SUMMARY:
The aim of the study is to develop an herbal gel based on Acmella oleracea and do a comparative analysis to evaluate the intensity of pain during the digital rectal examination comparing to lidocaine gel group and ultrasound gel group.

DETAILED DESCRIPTION:
The aim of the study is to develop an herbal gel based on Acmella oleracea and do a comparative analysis to evaluate the intensity of pain during the digital rectal examination comparing to lidocaine gel group and ultrasound gel group.

We are conducting a randomized, controlled, single-blind clinical trial of man undergoing to digital rectal examination, with 150 participants. Will be recruit at the Urologic Clinic of the Samuel Libânio Clinical Hospital and Urologic Clinic CISAMESP in Pouso Alegre. Participants divided into three groups, A. oleracea gel group, lidocaine gel group and ultrasound gel group. The digital rectal examination always performed by the same doctor, on the same position. A visual analogue scale (VAS) will be the standard method to evaluate the pain levels. The VAS will be explained to all patients, 0 = no pain and 10 = the most severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Patients to agree to participate in the study

Exclusion Criteria:

* Diabetic, chronic kidney disease, with urogenital infections, using an indwelling urinary catheter, with history of anorectal diseases or surgeries, psychiatric patients and who refused to participate in the research

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the pain | 1 day (After the digital rectal examination)
  A visual analogue scale (VAS) will be the standard method to evaluate the pain levels. The VAS will be explained to all patients, 0 = no pain and 10 = the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizia S Guerrieri, Principal Investigator — Vale do Sapucaí University
Locations (1):
- Universidade do Vale do Sapucaí, Pouso Alegre, Minas Gerais, Brazil